CLINICAL TRIAL: NCT05800106
Title: A Bioequivalence Study of Sunitinib Malate Capsules in Healthy Volunteers Under Fed Condition.
Brief Title: A Bioequivalence Study of Sunitinib Malate Capsules.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZDTQ-BE-2018-SNTN
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2018-08

CONDITIONS: Gastrointestinal Stromal Tumors; Renal Cell Carcinoma; Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Carcinoma, Renal Cell; Adenoma, Islet Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunitinib malate capsules generic product (Experimental): Single dose of Sunitinib malate capsule under fed condition on Day 1 and Day 29, respectively.
  Interventions: Drug: Sunitinib malate capsules generic product
- Sunitinib malate capsules reference product (Active Comparator): Single dose of Sunitinib malate capsule under fed condition on Day 1 and Day 29, respectively.
  Interventions: Drug: Sunitinib malate capsules reference product

INTERVENTIONS:
Drug: Sunitinib malate capsules generic product — Sunitinib is an inhibitor targeting multiple receptor tyrosine kinases (RTK).
  Arms: Sunitinib malate capsules generic product
Drug: Sunitinib malate capsules reference product — Sunitinib is an inhibitor targeting multiple receptor tyrosine kinases (RTK).
  Arms: Sunitinib malate capsules reference product

SUMMARY:
A randomized, open, two-period, two-sequence crossover trial design used to assess the pharmacokinetics and safety of Sunitinib Malate Capsules in healthy volunteers under fed condition, and compare the bioequivalence of Sunitinib Malate Capsules produced by Pfizer and Chia Tai Tianqing Pharmaceutical Group Co., Ltd, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent was signed before the study, fully understood the content and process of the study and the potential adverse reactions.
* Ability to complete the study in accordance with the protocol requirements.
* Chinese healthy adults aged 18-45 (included), male.
* Weight not less than 50 kg with a body mass index (BMI) between 18 and 28 kg/m2 (included, BMI = weight /height2).
* Health status: No mental abnormalities, no medical history of cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolic abnormalities.
* Vital signs, physical examination, laboratory examination, electrocardiogram and imaging examinations should be normal or abnormal with no clinical significance.
* Volunteers (including the partner) should ensure proper contraception from 2 weeks before dosing to at least 6 months after the last study drug administration, and ensure that one or more contraception measures are used in sexual during this period.

Exclusion Criteria:

* Previously suffered from neuropsychiatric system, respiratory system, cardiovascular system, gastrointestinal system, hemolymphatic system, liver and kidney insufficiency, endocrine system, musculoskeletal system diseases or other diseases, and the investigator judges that the past medical history may affect drug metabolism or safety.
* History of dysphagia or any gastrointestinal disorder affecting drug absorption.
* Have a history of intracranial hemorrhage or any disease that increases the risk of bleeding (such as repeated rhinorrhea, purpura, hemorrhoids, acute gastritis, etc.).
* Male subjects with clinically significant abnormal ECG history, or corrected QT (QTC) interval greater than 450 ms.
* People who have a history of dizziness of needles or blood.
* People who are allergic to sunitinib malate and its metabolites or its excipients.
* People who smoked more than 5 cigarettes per day in the 3 months before the clinical trial.
* People who have a history of drug and/or alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine).
* Blood donation or massive blood loss (> 450mL) within 2 months before taking study drug.
* Taking any drugs and contraceptives that change the activity of liver enzymes within 28 days before the study drug administration (such as liver drug enzyme inhibitors chlorpromazine, cimetidine, ciprofloxacin, metronidazole, etc.; liver drug enzyme inducers barbiturates, carbamazepine, rifampicin, dexamethasone, etc.).
* Taking any prescription drug, over-the-counter drug, any vitamin product, or herbal remedies within 14 days prior to the study drug administration.
* Need to use tobacco, alcohol and caffeinated drinks during the clinical trial, or certain foods that may affect metabolism (including dragon fruit, mango, grapefruit, and/or xanthine diet, etc.), or have significant changes in diet or exercise habits before the clinical trial , or other factors that affect drug absorption, distribution, metabolism, excretion, etc.
* Taking any study drug or participated in another drug clinical trial within 2 months before the study drug administration.
* Abnormal vital sign examination results with clinically significance.
* Abnormal clinical laboratory tests with clinically significance.
* Abnormal chest x-ray with clinically significance.
* Screening positive for hepatitis (including hepatitis B and C), Acquired immunodeficiency syndrome (AIDS), and syphilis.
* People who were positive in drug screening or had a history of drug abuse in the past five years or used drugs in the 3 months before the clinical trial.
* Difficulty or intolerance to blood collection by venipuncture.
* Acute illness occurred during the pre-study screening phase or prior to study medication.
* People who are unable to comply with ward management regulations.
* People who are unable to complete the clinical trial due to personal reasons.
* Other conditions that the investigator judges are not suitable for inclusion.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Maximum plasma concentration
Time to maximum concentration (Tmax) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Time to reach maximum concentration after drug administration
Area under the drug-time curve (AUC) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Area under the drug-time curve
Apparent terminal elimination half-life (t1/2) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Apparent terminal elimination half-life (t1/2)
Apparent volume of distribution (Vd/F) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Apparent volume of distribution
Clearance rate (CL/F) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Clearance rate
Apparent terminal elimination rate constant (λz) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Apparent terminal elimination rate constant
Relative bioavailability (F) | Before administration and 2, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96, 120, 168 hours after administration.
  Relative bioavailability (F) of the tested product to reference product

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  Incidence of adverse events (AE) evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) V5.0.
Severity of adverse events (AE) | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  Severity of adverse events (AE) evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal blood biochemistry results | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal blood biochemistry results evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal blood routine | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal blood routine results evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal urinalysis results | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal urinalysis results evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal coagulation function | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal coagulation function evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal thyroid function | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal thyroid function evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal blood pressure | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal blood pressure evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal pulse | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal pulse evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal body temperature | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal body temperature evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.
Proportion of subjects with abnormal 12-lead electrocardiogram (ECG) | From the date of randomization until the date of withdrawal from the study for any reason. Assessed up to 40 days.
  The proportion of subjects with abnormal 12-lead ECG evaluated in accordance with the National Cancer Institute's Common Toxicity Criteria (NCI CTC) v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China